CLINICAL TRIAL: NCT01917123
Title: Phase 0 Study of The Effect of L-Citrulline Malate on Ankle Brachial Index Among Patients With Coronary Heart Disease According to Their Smoking History
Brief Title: The Effect of L-Citrulline Malate on Ankle Brachial Index Among Patients With Coronary Heart Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Masih Daneshvari Hospital (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, babak sharif kashani, Head of Cardiology Department, Masih Daneshvari Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: f-91-128
Record Dates: First submitted 2013-08-03; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Heart Disease
Keywords: L-Citrulline malate,Coronary Heart Disease, Brachial Index
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimol, Brachial Index, Powder agent (Active Comparator): L-Citrulline malate,1gr,twice a day,2weeks
  Interventions: Drug: L-Citrulline malate
- Placebo, Brachial Index, Powder agent (Placebo Comparator): Placebo,1gr,twice a day,2weeks

INTERVENTIONS:
Drug: L-Citrulline malate — L-Citrulline malate as a 1gr powder agent, twice a day, for 2 weeks and placebo as a 1gr powder agent of O.R.S, twice a day,for 2 weeks
  Other Names: Stimol
  Arms: Stimol, Brachial Index, Powder agent

SUMMARY:
In this randomized clinical trial before and after study we will assess the effect of L-citrulline malate on brachial index in patients with coronary heart disease based on their smoking history. Twenty patients with coronary heart disease with no history of diabetes or other chronic diseases and with no history of myocardial infarction in the last 6 months will participate in our trial.A written well-versed permission was attained from all patients. We will measure the brachial index tow times once before giving L-Citrulline malate and the other time after 2 weeks giving it.Patients receiving L-Citrulline malate as a 1 gram dry powder agent twice a day, that should in use with 250 mg dilute water .The patients will followed after 2 weeks by measuring brachial index which is our primary outcome measurement in this trial.We assumed that the brachial index in both smoker and non-smoker group of patients with coronary heart disease would change to normal or close to normal after giving 1 gram L-citrulline malate twice a day for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1- patients with coronary heart disease without history of diabetes or any chronic disease 2- no myocardial infarction in last 6 months 3-ejection fraction more than 50% 4- please to recruit in the trial 5-no uncontrolled blood pressure 6- with stable condition when come to the clinic

Exclusion Criteria:

1- those who refuse to being in the trial 2- those which their total condition become worse 3- CCU admission as a result of being unstable 4- patients with chronic heart failure(CHF)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Brachial Index | 2 weeks
  Brachial Index according to the smoking history

SECONDARY OUTCOMES:
Brachial Index | 2 weeks
  Brachial Index according to coronary heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Babak Sharif-Kashani, Cardiologist, Study Director — Lung Transplantation Research Center, National Research Institute of Tuberculosis and Lung Diseases (NRITLD), Shahid Beheshti University of Medical Sciences, Tehran, Iran; Shabnam Eslam-Panah, M.D, Principal Investigator — Lung Transplantation Research Center, National Research Institute of Tuberculosis and Lung Diseases (NRITLD), Shahid Beheshti University of Medical Sciences, Tehran, Iran; Paritash Tahmaseb-pour, M.D, Principal Investigator — Lung Transplantation Research Center, National Research Institute of Tuberculosis and Lung Diseases (NRITLD), Shahid Beheshti University of Medical Sciences, Tehran, Iran
Locations (1):
- National Research Institute of Tuberculosis and Lung Diseases (NRITLD), Masih Daneshvari Hospital, Tehran, Tehran Province, Iran